CLINICAL TRIAL: NCT04818177
Title: Optimization of Dosing of Immunoglobulin G in the Obese Population
Brief Title: Immunoglobulin G Therapy Dose Optimization
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Luigi Brunetti, Associate Professor, Rutgers, The State University of New Jersey
Other Study IDs: Pro20160000739
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Immune Deficiency
Keywords: Pharmacokinetics; Obesity; Primary immune deficiency; Chronic inflammatory demyelinating polyneuropathy
MeSH Terms: conditions — Obesity; Immunologic Deficiency Syndromes; Primary Immunodeficiency Diseases; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

GROUPS / COHORTS (2):
- Normal Weight: Normal weight is defined as BMI 18.5 - 25 kg/m2. Subjects will receive the institutional standard intravenous immune globulin treatment.
  Interventions: Drug: Institutional standard intravenous immune globulin treatment
- Overweight or Obese: Overweight or obese is defined as BMI > 25 kg/m2. Subjects will receive the institutional standard intravenous immune globulin treatment.
  Interventions: Drug: Institutional standard intravenous immune globulin treatment

INTERVENTIONS:
Drug: Institutional standard intravenous immune globulin treatment — No treatments will be prospectively assigned. Subjects will receive their standard intravenous immune globulin doses. We will measure body composition and identify the relationship between body composition and intravenous immune globulin disposition.

SUMMARY:
The overall goal of this proposal is to investigate effects of obesity on pharmacokinetics of immunoglobulin G (IgG) and to develop strategies for optimization of dosing of IgG in obese patients. There is an ongoing debate regarding the most appropriate dosing of IgG formulations in obese patients. Obesity poses significant health risks; and evidence supporting dosing strategies of IgG in obese patients is inadequate. Some of the adverse reactions have been attributed to a relative overdosing in these patients, due to a limited distribution of IgG into fat tissue.

DETAILED DESCRIPTION:
The estimated prevalence of overweight and obese individuals >20 years in the US is 154.7 million (nearly double since the early 1960s), and over 1.6 billion people are considered overweight or obese worldwide. Compounding the health risks associated with obesity is the insufficient data supporting dosing strategies for a variety of medication used to treat conditions encountered in obese patients. No consensus on the best dosing strategy for IgG in obese patients has been established. Total (TBW), ideal (IBW), and adjusted (AdjBW) body weight-based dosing are being utilized by different institutions. Thus, there is an urgent need to identify evidence supporting optimal dosing strategies for IgG.

It has been proposed that using TBW to dose IgG in obese patients may increase the risk of thrombosis owing to increased blood viscosity, activation of platelets, or vasospasm; and the increase in blood viscosity has been reported as IgG dose dependent. The use of using IBW or AdjBW has been advocated to reduce the side effect and drug expenditures. It is currently unknown what the clinical impact is of using measures of body weight other than TBW to calculate IgG doses, and the effect of obesity on IgG pharmacokinetics has not been experimentally evaluated.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 75 years
* currently treated with IVIG

Exclusion Criteria:

* liver impairment (elevations in liver enzymes of greater than 3 times the upper limit of normal)
* reduced renal function (CrCl < 50 mL/min)
* Patients with a pacemaker or an automatic implantable cardioverter-defibrillator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients receiving the institutional standard intravenous immune globulin therapy. Differences in IgG concentrations will be analyzed between normal weight subjects (BMI 18.5 - 25 kg/m2) and overweight or obese subjects (BMI > 25 kg/m2).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum IgG concentrations | 5 time points (baseline, immediately after dose administration (peak), 2 weeks post dose, just prior to receiving the next scheduled dose (trough))
  A linear mixed effects model to analyze serum IgG concentrations, with normal/obese as the primary predictor but with clinical and demographic variables as covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Brunetti, Ph D; PharmD, Principal Investigator — Rutgers University
Locations (1):
- Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No